CLINICAL TRIAL: NCT05809544
Title: A Randomized, Double-blinded, Sham-controlled Clinical Trial to Evaluate the Safety and Efficacy of Digital Cognitive Behavioral Therapy for Insomnia
Brief Title: Study of Efficacy of WELT-IP in Insomnia (WCTP-I-B-02)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WELT corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WCTP-I-B-02
Record Dates: First submitted 2023-03-13; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Insomnia
Keywords: digital therapeutics
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded design, with three points of measurement. The subjects will receive either the WELT-IP app or sham app.
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WELT-IP (Experimental): Eligible subjects were able to access WELT-IP (an investigational digital therapeutic) on a mobile device (iOS and Android) as scheduled to receive CBT-I.
  Interventions: Device: WELT-IP
- Sham (Sham Comparator): Eligible subjects were able to access a sham app downloaded on a mobile device (iOS and Android) which included sleep diary and general content regarding sleep.
  Interventions: Device: Sham

INTERVENTIONS:
Device: WELT-IP — WELT-IP (an investigational digital therapeutic) is an CBT-I based intervention designed to treat insomnia, conducted in 6 sessions. It is a comprehensive program delivering sleep restriction, stimulation control, muscle relaxation, cognitive treatment, and sleep hygiene education. Main features are sleep diary, sleep reports, daily lessons of CBT-I, muscle relaxation techniques, and cognitive intervention through chatbot.
  Arms: WELT-IP
Device: Sham — Sham was downloaded to the subject's phone and was subject was instructed to complete sleep diary and sleep educational contents as needed.
  Arms: Sham

SUMMARY:
The purpose of the study was to determine safety and efficacy of WELT-IP in adult insomnia patients. WELT-IP is a cognitive behavioral therapy for insomnia (CBT-I) based digital therapeutics.

DETAILED DESCRIPTION:
This was a randomized, double-blinded, sham-controlled trial. Overall, 68 subjects were randomized into the following groups:

* WELT-IP group: WELT-IP (insomnia digital therapeutics) use
* Control group: sham app use Subjects in both groups continued to receive their clinician-directed standard-of-care treatment for insomnia, if applicable, including pharmacotherapy. After screening of sleep diary, subjects were randomized and in WELT-IP group used WELT-IP and subjects in control group used a sham for a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 insomnia patient
* SE (sleep efficiency) <80%
* completing screening sleep diary of 7 consecutive days
* ISI of 8 or above
* capable of using mobile device and application

Exclusion Criteria:

* currently on non-pharmacological treatment for insomnia (ex. CBT-I, light therapy, oriental therapy for insomnia)
* sleep disorders diagnosis other than insomnia (ex. Obstructive sleep apnea, sleep behavior problem, restless leg syndrome)
* progressive and active medical conditions
* received continuous psychotherapy such as CBT, motivational enhancement therapy, psychotherapy, and psychoanalysis in the past 3 months
* major psychiatric illness as assessed through MINI
* suicide risk as assessed through C-SSRS
* having occupational risk due to sleep restriction
* shift workers

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 7 (post-treatment) of Sleep efficiency(SE) | 7 weeks
  Sleep efficiency is calculated as percentage of Total sleep time/Time in bed.

SECONDARY OUTCOMES:
Change from baseline to week 7 (post-treatment) of Sleep quality (SQ) | 7 weeks
  Sleep quality ranges from 1 to 5, where higher score indicates better quality of sleep.
Change from baseline to week 7 (post-treatment) of Sleep onset latency (SOL) | 7 weeks
  Sleep onset latency is evaluated as the time it takes a person to fall asleep after going to bed.
Change from baseline to week 7 (post-treatment) of Wake after sleep onset (WASO) | 7 weeks
  Wake after sleep onset is calculated as the total number of minutes that a person is awake after initially falling asleep.
Change from baseline to week 7 (post-treatment) of Total sleep time (TST) | 7 weeks
  Total sleep time is calculated as the total number of minutes that a person actually sleep.
Change from baseline to week 7 (post-treatment) of Number of awakening (NOA) | 7 weeks
  Number of awakening is evaluated as the number of times a person wakes up after falling asleep.
Change from baseline to week 7 (post-treatment) of Insomnia severity index (ISI) | 7 weeks
  Insomnia severity index has seven questions. Total score ranges from 0 to 28, where higher scores indicate more acute symptoms of insomnia.
Change from baseline to week 7 (post-treatment) of Dysfunctional beliefs and attitudes about sleep-16 (DBAS-16) | 7 weeks
  Dysfunctional beliefs and attitudes about sleep-16 has sixteen questions. Responses can range from 0 to 10, where higher scores indicate more irrational beliefs and attitudes toward sleep.
Change from baseline to week 7 (post-treatment) of Patient health questionnaire-9 (PHQ-9) | 7 weeks
  Patient health questionnaire-9 has nine questions. Total score ranges from 0 to 27, where higher scores indicate more acute symptoms of depression.
Change from baseline to week 7 (post-treatment) of Generalized anxiety disorder-7 item scale (GAD-7) | 7 weeks
  Generalized anxiety disorder-7 item scale has seven questions. Total score ranges from 0 to 21, where higher scores indicate more acute symptoms of anxiety.
Percentage of subjects achieving SE ≥ 85% | 7 weeks
Compliance (completion rate of lessons, for WELT-IP group only) | 7 weeks
  Compliance is evaluated as completion rate of lessons.

OTHER OUTCOMES:
App Satisfaction Survey | 7 weeks
Sleep Environment Survey | 7 weeks
Activity data from mobile device | 7 weeks
  Activity data is evaluated as change of number of steps from baseline to week 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Park KM, Lee DH, Choi EC, Lee Y, Lee E. Impact of Adherence to Digital Cognitive Behavioral Therapy for Insomnia Effectiveness. Yonsei Med J. 2025 Oct;66(10):657-665. doi: 10.3349/ymj.2024.0398. PMID 40992766